CLINICAL TRIAL: NCT02233907
Title: Post-marketing Surveillance (as Per § 67(6) AMG [German Drug Law]) of Ventilat® in Long-term Therapy in Chronic Obstructive Pulmonary Disease
Brief Title: Post-marketing Surveillance of Ventilat® in Long-term Therapy in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 54.563
Record Dates: First submitted 2014-09-08; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease patients
  Interventions: Drug: Ventilat® - metered dose inhaler

INTERVENTIONS:
Drug: Ventilat® - metered dose inhaler

SUMMARY:
Study to obtain further information on the tolerability and efficacy of Ventilat® metered dose inhaler in long-term treatment of Chronic Obstructive Pulmonary Disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders older than 40 years, who suffer from Chronic Obstructive Pulmonary Disease
* Only patients who have not been treated with Ventilat® within the last year are to be considered for inclusion

Exclusion Criteria:

* Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Ventilat® metered dose inhaler

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic obstructive pulmonary disease at general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 1999-10; Primary Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Change in the clinical picture | up to 12 months

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | after 12 months
Assessment of efficacy by patient on a 4-point scale | after 12 months
Number of patients with adverse drug reactions | up to 12 months
Assessment of tolerability by investigator on a 4-point scale | after 12 months
Assessment of tolerability by patient on a 4-point scale | after 12 months